CLINICAL TRIAL: NCT02438150
Title: The Effectiveness of an On-line Training Program on Hospital Medical Staff to Improve Fire Knowledge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Paul Lee, Research Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: HSEARS20141020002
Record Dates: First submitted 2015-04-27; First posted 2015-05-08 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Fire
Keywords: Disaster; Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Will receive hospital fire video training
  Interventions: Behavioral: Hospital fire video training
- Control (Placebo Comparator): Will receive non-fire video training
  Interventions: Behavioral: Non hospital fire video training

INTERVENTIONS:
Behavioral: Hospital fire video training — Participants will watch a video about hospital fire training which last for 30 minutes
  Arms: Intervention
Behavioral: Non hospital fire video training — Participants will watch a video about volcanic eruption which last for 30 minutes
  Arms: Control

SUMMARY:
Objective: To investigate the effectiveness of an online training program on medical staff in five public hospitals located in Sichuan, Yunnan, Hubei, and Fujian Provinces of China, on improving fire knowledge.

Methods: Participants will be randomly divided into control (receiving non-fire video training) and intervention (receiving hospital fire video training) groups. All participants will complete a questionnaire of fire knowledge before and after receiving the training.

Hypothesis: If the online training is effective, it can be promoted as a convenient and effective use of training and be promoted to other hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Physicians or nurses working in the recruiting hospitals

Exclusion Criteria:

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2015-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change of fire knowledge | Participants will complete the questionnaire 5 minutes before the start of and 1 minute after watching the video which last for 30 minutes, and the change of fire knowledge will be computed.
  A 46-item multiple-choice questionnaire will be administered to measure the fire knowledge level of the participants. Sample items include "Use a wet towel to cover your nose and mouth when fire occurs" and "How to assist patients with intravenous infusion to escape?".

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Hospital, Chengdu, Sichuan, China

REFERENCES:
- [Derived] Lee PH, Fu B, Cai W, Chen J, Yuan Z, Zhang L, Ying X. The effectiveness of an on-line training program for improving knowledge of fire prevention and evacuation of healthcare workers: A randomized controlled trial. PLoS One. 2018 Jul 5;13(7):e0199747. doi: 10.1371/journal.pone.0199747. eCollection 2018. PMID 29975723